CLINICAL TRIAL: NCT03633942
Title: Safety and Efficacy of the LMA Supreme Supraglottic Airway Device When Used for Adult Patients Undergoing Spinal Surgery in the Prone Position
Brief Title: Safety and Efficacy of the LMA Supreme When Inserted With Patients in the Prone Position
Acronym: LMA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Laser Spine Institute (Industry)
Collaborators: Teleflex (Industry)
Responsible Party: Sponsor
Other Study IDs: LMA 200
Record Dates: First submitted 2018-06-29; First posted 2018-08-16 (Actual); Last update posted 2018-08-24 (Actual); Status verified 2018-08

CONDITIONS: Airway Obstruction
MeSH Terms: conditions — Airway Obstruction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Observational: LMA Supreme: An appropriately sized LMA Supreme will be prepared by removing all air from the cuff while applying manual pressure. A water soluble non-local anesthetic containing lubricant gel will be applied to the fully deflated airway before insertion. A 1 cm column of the gel will be preloaded into the gastric port of the LMA Supreme for the Gel Test.
  The cuff will be inflated with a manometer to a pressure of approximately 30cm H2O. If a significant leak is detected, the cuff will be inflated in increments of 5cm H2O until a satisfactory seal is obtained. The final cuff pressure will be recorded. The lungs will then be gently inflated by applying manual pressure to the anesthesia circuit bag while observing the gel column in the LMA Supreme gastric port for movement.
  Interventions: Device: LMA Supreme

INTERVENTIONS:
Device: LMA Supreme — Placement of the LMA Supreme supraglottic airway device for patients undergoing outpatient spine surgery in the prone position.

SUMMARY:
This study is a non-randomized, observational, non-comparative prospective study to evaluate the safety, efficacy and performance of the LMA Supreme laryngeal mask airway when used according to the device's Instructions for Use.

DETAILED DESCRIPTION:
This study is a non-randomized, observational, non-comparative prospective study to evaluate the safety, efficacy and performance of the LMA Supreme laryngeal mask airway when used according to the device's Instructions for Use. During surgery, standard treatment will be applied, complemented with the recording of study parameters related to safety, efficacy and performance of the LMA Supreme laryngeal mask airway.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 70 years of age
* American Society of Anesthesiology Classification (ASA) I-III patients
* Fasting for 8 hours
* Scheduled surgery with indication for laryngeal mask airway

Exclusion Criteria:

* Have contraindicating conditions
* Have had radiotherapy to the neck involving the hypopharynx (risk of trauma, failure to seal effectively).
* Have inadequate mouth opening to permit insertion
* History of hiatal hernia
* Scheduled for minimally invasive spine stabilization procedures such as Transforaminal Lumbar Interbody Fusion (TLIF), Anterior Cervical Discectomy and Fusion (ACDF) (all have neuromonitoring/general endotracheal intubation)
* Scheduled for Joimax procedure (initial anesthetic is MAC)
* Unable to safely position themselves prone with assistance
* History of previous failed LMA Supreme placement
* BMI greater than or equal to 53
* Outside age or ASA range specified in inclusion criteria
* Inability to comply with study requirements including follow-up

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients undergoing outpatient spine surgery in the prone position that meet the eligibility criteria.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2018-07-27 (Actual); Primary Completion 2019-07-27 (Estimated); Study Completion 2020-07-27 (Estimated)

PRIMARY OUTCOMES:
The efficacy of the LMA Supreme device as assessed by measurement of ventilation on Case Report Form 1 | Intraoperative
  Outcome being measured intraoperatively is the ease of manual ventilation via the LMA Supreme. Measuring, no air leaks, air leak / elevated airway pressure needed for adequate ventilation, removal and reinsertion needed to achieve adequate ventilation, no ventilation after 2 attempts (airway managed using alternative techniques
The efficacy of the LMA Supreme device as assessed by measurement of ease of swallowing on Case Report Form 2 | Preoperative and up to 4 weeks (+/- 5 days) postoperative
  Outcome being measured preoperatively and at 4 weeks +/- 5 days is the Dysphagia (difficulty swallowing) Short Questionnaire. Measuring the ability to swallow (any difficulty in swallowing), incorrect swallowing (any coughing associated with swallowing), lump feeling (any lumps in the throat), involuntary loss of weight (any weight loss recently), Pneumonia (any bouts with pneumonia).
The efficacy of the LMA Supreme device as assessed by measurement of removal of the LMA Supreme Device on Case Report Form 1 | Intraoperative
  Outcome being measured intraoperatively is any blood on the LMA upon removal. Measuring if there is minimal or no blood, blood covering less than one fourth of the LMA or blood on at least one half of the LMA surface.
The efficacy of the LMA Supreme device as assessed by measurement of any intraoperative episodes developing reporting outcomes on Case Report Form 1 | Intraoperative
  Outcome being measured intraoperatively is did patient develop any intraoperative episodes of laryngospasm, hiccups, or coughing.

SECONDARY OUTCOMES:
Dysphagia Short Questionnaire | Preoperative and up to 4 weeks postoperative (+/- 5 days).
  Instrument used to measure difficulty swallowing (dysphagia).

CONTACTS AND LOCATIONS:
Overall Officials: Thor Van Diver, MD, Principal Investigator — Laser Spine Institute; George Lin, MD, Principal Investigator — Laser Spine Institute
Locations (1):
- Laser Spine Institute, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Smith I, White PF. Use of the laryngeal mask airway as an alternative to a face mask during outpatient arthroscopy. Anesthesiology. 1992 Nov;77(5):850-5. doi: 10.1097/00000542-199211000-00003. PMID 1443736
- [Background] Brimacombe J. The advantages of the LMA over the tracheal tube or facemask: a meta-analysis. Can J Anaesth. 1995 Nov;42(11):1017-23. doi: 10.1007/BF03011075. PMID 8590490
- [Background] Brimacombe JR, Berry A. The incidence of aspiration associated with the laryngeal mask airway: a meta-analysis of published literature. J Clin Anesth. 1995 Jun;7(4):297-305. doi: 10.1016/0952-8180(95)00026-e. PMID 7546756
- [Background] Joshi GP, Inagaki Y, White PF, Taylor-Kennedy L, Wat LI, Gevirtz C, McCraney JM, McCulloch DA. Use of the laryngeal mask airway as an alternative to the tracheal tube during ambulatory anesthesia. Anesth Analg. 1997 Sep;85(3):573-7. doi: 10.1097/00000539-199709000-00016. PMID 9296411
- [Background] Koga K, Asai T, Vaughan RS, Latto IP. Respiratory complications associated with tracheal extubation. Timing of tracheal extubation and use of the laryngeal mask during emergence from anaesthesia. Anaesthesia. 1998 Jun;53(6):540-4. doi: 10.1046/j.1365-2044.1998.00397.x. PMID 9709138
- [Background] Hohlrieder M, Brimacombe J, Eschertzhuber S, Ulmer H, Keller C. A study of airway management using the ProSeal LMA laryngeal mask airway compared with the tracheal tube on postoperative analgesia requirements following gynaecological laparoscopic surgery. Anaesthesia. 2007 Sep;62(9):913-8. doi: 10.1111/j.1365-2044.2007.05142.x. PMID 17697218
- [Background] van Zundert A, Brimacombe J. The LMA Supreme--a pilot study. Anaesthesia. 2008 Feb;63(2):209-10. doi: 10.1111/j.1365-2044.2007.05421.x. No abstract available. PMID 18211462
- [Background] Verghese C, Ramaswamy B. LMA-Supreme--a new single-use LMA with gastric access: a report on its clinical efficacy. Br J Anaesth. 2008 Sep;101(3):405-10. doi: 10.1093/bja/aen174. Epub 2008 Jun 17. PMID 18559351
- [Background] Truhlar A, Ferson DZ. Use of the Laryngeal Mask Airway Supreme in pre-hospital difficult airway management. Resuscitation. 2008 Aug;78(2):107-8. doi: 10.1016/j.resuscitation.2008.03.008. Epub 2008 May 27. No abstract available. PMID 18508181
- [Background] Edgcombe H, Carter K, Yarrow S. Anaesthesia in the prone position. Br J Anaesth. 2008 Feb;100(2):165-83. doi: 10.1093/bja/aem380. PMID 18211991
- [Background] Sharma V, Verghese C, McKenna PJ. Prospective audit on the use of the LMA-Supreme for airway management of adult patients undergoing elective orthopaedic surgery in prone position. Br J Anaesth. 2010 Aug;105(2):228-32. doi: 10.1093/bja/aeq118. Epub 2010 Jun 10. PMID 20542887
- [Background] [The Helsinki Declaration of the World Medical Association (WMA). Ethical principles of medical research involving human subjects]. Pol Merkur Lekarski. 2014 May;36(215):298-301. No abstract available. Polish. PMID 24964504